CLINICAL TRIAL: NCT03504228
Title: Prospective, Single-arm, Multi-center, Observational Study to Further Confirm Safety and Efficacy of the Dual-layer Micromesh Roadsaver Stent for the Treatment of Carotid Artery Stenosis in Patients Eligible for Elective Stenting Procedure
Brief Title: Prospective Single Arm CAS - ROADSAVER Study
Acronym: ROADSAVER
Status: Completed | Type: Observational
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: T130E2
Record Dates: First submitted 2018-03-15; First posted 2018-04-20 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-01

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Roadsaver — Dual layer micromesh Roadsaver carotid stent

SUMMARY:
Approximately 2000 patients eligible for elective treatment with a Carotid Stent according to hospital routine practice in centers across Europe will be enrolled in the study. The maximum number of patients enrolled at each site will be not limited. Follow-ups are scheduled at discharge, 30 days, and 1 year, as per local practice. Each patient will have follow-up contacts via hospital visit and/or telephone.

DETAILED DESCRIPTION:
1. Baseline Assessments

   The patient will be assessed in accordance with the hospital standard of care for patients treated with carotid artery stenting procedure, which in general includes:
   * Informed consent for data collection
   * Demographics
   * Medical History
   * Medication record
   * Physical examination
   * Carotid Duplex Ultrasound
   * Neurological Assessment
   * Diffusion weighted Magnetic Resonance Imaging (DW-MRI)
   * Procedural angiography

   Baseline assessments will be performed prior to the index procedure and documented in the patient medical record. Baseline assessments considered standard of care completed prior to obtaining informed consent do not need to be repeated unless the investigator feels it is medically necessary.

   Neurological Assessment Baseline neurological assessment is recommended in this study and will be conducted by a physician, nurse, or other allied health professional, independent of the treating physician prior to the procedure. This assessment will include the neurological signs, symptoms, and the NIH Stroke Scale. For some pre-specified subgroups, imaging studies (Carotid Duplex Ultrasound and/or Diffusion Weighted Magnetic Resonance Imaging: DW-MRI) will be performed prior to the procedure.
2. Patient Enrollment Point A patient is considered enrolled in the study if there is full compliance with the study and RoadSaver IFU eligibility criteria, and only after successful guidewire passage through the study target lesion.
3. Medications Patients enrolled in this study will be pre-medicated according to the hospital routine practice.
4. Procedure The procedure will be performed according to the physician's standard of care. During the procedure, patients should receive appropriate anticoagulation and other therapy according to standard hospital practice. The use of any medication for the treatment of vessel spasm, patient agitation or discomfort, hypotension, arrhythmias, and hemodynamic changes during the procedure is at the discretion of the investigator.

   Standard procedures should be followed based on the Instructions for Use for the Roadsaver™ device of Terumo. If pre- and/or post-dilatation is performed, or any other device (e.g. embolic protection devices, etc.) is used at the investigator's discretion.

   4.1. Treatment Failures If a Roadsaver™ Carotid Stent is not implanted due to technical reasons, another CE-marked Carotid Stent may be used to complete the procedure. Patients who do not have a successful Roadsaver™ Carotid Stent implanted during the index procedure will be considered as technical failures.

   Patients with technical failure will be followed only until discharge at which time they will have completed the study.

   All patients who receive a Roadsaver™ Carotid Stent upon enrollment in the ROADSAVER study will be included in the analysis of clinical outcomes by the end of the study. Patients with technical failures will be analyzed separately only for procedural success and for in-hospital adverse events.

   4.2. Device Deficiency and Device Malfunction A device deficiency is defined as an inadequacy of a medical device related to its identity, quality, durability, reliability, safety, or performance. This may include malfunctions, use error, or inadequacy in the information supplied by the manufacturer.

   A device malfunction is defined as failure of the medical device to perform in accordance with its intended purpose when used in accordance with the instructions for use or the Clinical Investigation Plan.

   In case of device deficiency or malfunction, the device deficiency form in the eCRF should be completed and the investigator is asked to make every possible effort to return the device to Terumo Europe accompanied if possible with the packaging containing the device identification (lot number). Another Roadsaver™ Carotid Stent or another stent as per operators' discretion will be used in order to complete the treatment of the patient.
5. Post-procedure

   Post-procedural evaluation should be done according to the routine hospital practice prior to discharge, which in general includes:
   * Post Angiography immediately after the index procedure
   * Physical examination before discharge
   * MAE defined as the cumulative incidence of any periprocedural death or stroke
   * Adverse events including: any revascularization, major vascular and bleeding complications, other
   * Medication
   * Neurological assessment when performed
   * Diffusion-weighted magnetic resonance imaging (DW-MRI) when performed

   Information on the post-procedural evaluation and any interventional treatment that occurred since the procedure should be collected.
6. Follow-Up Evaluations Patients will be followed according to routine hospital practice usually performed at 30-day and at 12-month assessment through hospital visit or through telephone contact. Investigators and research coordinators will keep notes of all telephone contacts with the patients in the patient hospital file as source documents.

Hospital Visit at 1 month (30 ± 7 days) and 12 months (365 ± 30 days) Patients' clinical status should be reported if hospital visits are done at 30 days and 12 months.

These follow-up assessments should be done according to the routine hospital practice, which in general includes:

* Physical examination
* Adverse events including: any stroke, any Revascularization, major vascular and bleeding complications, other
* Medication
* Neurological assessment
* Carotid duplex ultrasound
* Diffusion-weighted magnetic resonance imaging (DW-MRI)

All relevant information obtained during follow-up including imaging should be reported. Data to be collected at follow-ups would include:

Telephone Contact at 12 months (365 ±30 days)

* Adverse Events including: any death (stroke related/other), any stroke, any revascularization, major vascular and bleeding complications, other
* Medication In case of death, stroke, TLR, and TVR all efforts should be made to provide sufficient baseline and event documentation.

Unscheduled Follow-Up

The assessment at unscheduled visits should be performed according to safety reporting requirements, which in general includes:

* Physical examination
* Adverse events including: any stroke, any revascularization, major vascular and bleeding complications, other
* Medication
* Neurological assessment
* Carotid duplex ultrasound
* Diffusion-weighted magnetic resonance imaging (DW-MRI)

A patient who returns to the investigational site between pre-determined visits with an event related to the index procedure should be treated according to the physician's standard of care. Reportable events occurring during this period should be collected.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a non-occlusive and non-thrombotic carotid artery stenosis and is eligible to be treated with Roadsaver Carotid Stent as per the Instructions for Use (IFU)
* The patient is at least 18 years of age
* The patient has a life expectancy of at least 12 months from the date of the index procedure
* The patient is able and willing to provide a signed IRB-/EC-approved informed consent form prior to participation

Exclusion Criteria:

- Any condition that makes patient unsuitable for percutaneous transluminal angioplasty (PTA), including intolerance or allergy to any material used and accompanying therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in this study will be comprised of male and female patients derived from general interventional radiology or angiology populations.
Sampling Method: Probability Sample
Enrollment: 1967 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
The rate of Major Adverse Events (MAE) | Up to 30 days
  Defined as the cumulative incidence of any death or stroke up to 30 days after the index procedure.

SECONDARY OUTCOMES:
Technical Success | Peri-procedural
  Defined as a successful access and deployment of the device with recanalization, determined by <30% residual stenosis by angiography during the index procedure.
Procedural success | Peri-procedural
  Defined as technical success with no device-/procedure-related death, stroke or any other serious adverse events.
Device malfunction | Peri-procedural
  Defined as the failure of a device after its introduction into the patient (i.e. failure to perform in accordance with its intended purpose when used as per the Instructions For Use or the Clinical Investigation Plan).
Any death | Up to 30 days
  Adjudicated by an independent Clinical Events Committee.
Stroke-related death | Up to 30 days
  Defined as a death which has been adjudicated by an independent clinical events committee to have directly resulted from a stroke.
Any stroke | Up to 30 days
  Defined as an acute neurologic event with focal symptoms and signs, lasting for 24 hours or more (Adjudicated by an independent Clinical Events Committee).
Major stroke | Up to 30 days
  Defined as a new neurological event that persists for > 24 hours and results in a > 4 point increase in the NIHSS score relative to baseline or any subsequent lower score (Adjudicated by an independent Clinical Events Committee).
Minor stroke | Up to 30 days
  Defined as a new neurological event that resolves completely within 7 days or increases the NIHSS by ≤4 points (Adjudicated by an independent Clinical Events Committee).
Transient ischemic attack | Up to 30 days
  TIA
Target lesion revascularization (TLR) | Up to 30 days
  Defined as any revascularization procedure of the original treatment site, including angioplasty, stenting, endarterectomy, or thrombolysis, performed to open or increase the luminal diameter inside or within 5 mm of the previously treated lesion (Adjudicated by an independent clinical events committee).
Major vascular and bleeding complications: | Up to 30 days
  1. Major hematoma, i.e. one requiring transfusion, surgical evacuation, or delay in discharge,
  2. Pseudo aneurysm or arteriovenous fistula or retroperitoneal bleeding,
  3. Peripheral ischemia/nerve injury caused by the proximal access site,
  4. Vascular surgical repair to correct a local vascular access site complication and bleeding.

OTHER OUTCOMES:
Any death (Rate assessed in a subgroup of patients that undergoes 12-month follow-up as per standard of care) | Up to 12 months
  Adjudicated by an independent Clinical Events Committee.
Stroke-related death (Rate assessed in a subgroup of patients that undergoes 12-month follow-up as per standard of care) | Up to 12 months
  Adjudicated by an independent Clinical Events Committee.
Any stroke (Rate assessed in a subgroup of patients that undergoes 12-month follow-up as per standard of care) | Up to 12 months
  Defined as an acute neurologic event with focal symptoms and signs, lasting for 24 hours or more, adjudicated by an independent Clinical Events Committee.
Ipsilateral stroke (Rate assessed in a subgroup of patients that undergoes 12-month follow-up as per standard of care) | Up to 12 months
  Defined as a stroke occurring within the vascular distribution of the stented artery, adjudicated by an independent Clinical Events Committee.
Target lesion revascularization (Rate assessed in a subgroup of patients that undergoes 12-month follow-up as per standard of care) | Up to 12 months
  Defined as any revascularization procedure of the original treatment site, including angioplasty, stenting, endarterectomy, or thrombolysis, performed to open or increase the luminal diameter inside or within 5 mm of the previously treated lesion (Adjudicated by an independent clinical events committee).
In-stent restenosis (Rate assessed in a subgroup of patients that undergoes 12-month follow-up as per standard of care) | Up to 12 months
  Measured within the stented lesion or within 5 mm proximal or distal to the stent, defined as ≥50% stenosis by ultrasound (Peak Systolic Velocity Ratio (PSVR; PSV(ICA) / PSV(CCA) >2) or ≥ 70% stenosis by angiography).
External carotid artery patency (Rate assessed in a subgroup of patients that undergoes 12-month follow-up as per standard of care) | Up to 12 months
  Determined as per ultrasound assessment

CONTACTS AND LOCATIONS:
Overall Officials: Ihsen Merioua, MD, Study Director — Ihsen.Merioua@terumo-europe.com
Locations (57):
- Belgium (5):
  - OLV Ziekenhuis, Aalst
  - Imelda Ziekenhuis, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
- Czechia (2):
  - University Hospital Ostrava, Ostrava
  - Central Military Hospital Prague, Prague
- France (4):
  - GCS Centre de Cardiologie du Pays Basque, Bayonne
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Hopital de la Timone 2, Marseille
  - Polyclinique Louis Pasteur Essey Les Nancy, Nancy
- Germany (13):
  - Ihre-Radiologen.de, Berlin
  - Sankt-Gertrauden Krankenhaus, Berlin
  - Fürst-Stirum-Klinik, Bruchsal
  - Diakonissenkrankenhaus Flensburg Ev.-Luth. Diakonissenanstalt zu Flensburg, Flensburg
  - Cardioangiological Center Bethanien, Frankfurt am Main
  - SRK Karlsbad, Karlsbad
  - Theresienkrankenhaus Mannheim, Mannheim
  - St. Franziskus-Hospital Münster, Münster
  - Pius Hospital Oldenburg, Oldenburg
  - Klinikum Passau, Passau
  - Elblandklinikum Radebeul, Radebeul
  - SRH Zentralklinikum Suhl, Suhl
  - Universitäts und Rehabilitationskliniken Ulm, Ulm
- Hungary (7):
  - Markusovszky Teaching Hospital, Budapest
  - Semmelweis University Heart and Vascular Center, Budapest
  - Moritz Kaposi Teaching Hospital, Kaposvár
  - Bacs-Kiskun County Hospital, Kecskemét
  - University of Pécs, Pécs
  - Szeged University Hospital, Szeged
  - Szent György Fejér County - University Teaching Hospital, Székesfehérvár
- Paul Stradins Clinical University Hospital, Riga, Latvia
- Netherlands (2):
  - UMC Groningen, Groningen
  - Sint-Antonius Ziekenhuis, Nieuwegein
- North Macedonia (2):
  - City General Hospital 8th September Skopje, Skopje
  - University Clinic of Cardiology, Skopje
- Poland (3):
  - Szpital Uniwersytecki nr.2 im. Dr J. Biziela w Bydgoszczy, Bydgoszcz
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow
  - Szpital Uniwersytecki w Krakowie, Krakow
- Centro Hospitalar Vilanova Gaia/Espinho, Vila Nova de Gaia, Portugal
- Serbia (3):
  - Clinical Center of Serbia, Belgrade
  - ICVD Dedinje, Belgrade
  - Clinical Center of Vojvodina, Novi Sad
- Slovakia (2):
  - Cinre S.R.O., Bratislava
  - Kardiocentrum Nitra, Nitra
- Spain (12):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Clinico de Barcelona, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Hospital Universitario Girona Josep Trueta, Girona
  - Complejo Hospitalario De Jaen, Jaén
  - Hospital 12 de Octubre, Madrid
  - Hospital Quironsalud Marbella, Marbella
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario Donostia, San Sebastián
  - Hospital universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Virgen de La Salud de Toledo, Toledo
  - Hospital Universitario Clínico de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muller-Hulsbeck S, Vajda Z, Odrowaz-Pieniazek P, Ruzsa Z, Beelen R, Gjoreski A, Deloose K, Castro S, Faurie B, Tomasello Weitz A, Schwindt A, Latacz P, Orgaz Perez-Grueso A, Cvetic V, Langhoff R, Kedev S; all ROADSAVER study investigators. Contemporary carotid artery stenting practices and peri-procedural outcomes in different European countries: ROADSAVER study multicentric insights. CVIR Endovasc. 2025 Apr 12;8(1):29. doi: 10.1186/s42155-025-00528-z. PMID 40220262
- [Derived] Kedev S, Muller-Hulsbeck S, Langhoff R. "Real-World Study of a Dual-Layer Micromesh Stent in Elective Treatment of Symptomatic and Asymptomatic Carotid Artery Stenosis (ROADSAVER)". Cardiovasc Intervent Radiol. 2022 Mar;45(3):277-282. doi: 10.1007/s00270-021-03051-5. Epub 2022 Jan 18. PMID 35043241